CLINICAL TRIAL: NCT00084903
Title: Pathological Correlation of Colposcopically Directed Biopsies to Fluorescence EEM of the Normal Human Cervix
Brief Title: Fluorescence and Reflectance Spectroscopy During Colposcopy in Detecting Cervical Intraepithelial Neoplasia and Dysplasia in Healthy Participants With a History of Normal Pap Smears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GYN97-244; P30CA016672 (NIH); MDA-GYN-97244 (Other: UT MD Anderson Cancer Center); UTHSC-HSC-MS-04-307; BCCA-RO2-1476; CDR0000366944 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Biopsy; Spectrum Analysis; Spectrometry, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluorescence Spectroscopy (Experimental)
  Interventions: Procedure: Colposcopic biopsy; Procedure: Light-Scattering Spectroscopy

INTERVENTIONS:
Procedure: Colposcopic biopsy — Two small samples of cervical tissue (biopsy) removed from 2 sites as spectroscopy readings.
  Other Names: biopsy
Procedure: Light-Scattering Spectroscopy — Spectroscopy readings taken in 2 regions of cervix.
  Other Names: Spectroscopy; Fluorescence spectroscopy

SUMMARY:
RATIONALE: New diagnostic procedures such as fluorescence and reflectance spectroscopy (shining light on tissue and measuring patterns of light reflected) may improve the ability to noninvasively detect cervical intraepithelial neoplasia and dysplasia.

PURPOSE: This diagnostic trial is studying how well fluorescence and reflectance spectroscopy during colposcopy work in detecting cervical intraepithelial neoplasia and dysplasia in healthy participants with a history of normal Pap smears.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify potential improvements in noninvasive methods of diagnosing dysplasia and neoplasia of the cervix using fluorescence and reflectance spectroscopy in healthy participants with a history of normal pap smears.
* Determine the reflection and fluorescence spectra of in vivo samples of the normal human cervix.
* Refine the detection of cervical lesions by fluorescence spectroscopy in these participants using improved classification of normal columnar tissue and non-neoplastic tissue with inflammation.
* Determine and validate the wavelength selections for spectroscopic diagnosis derived from in vitro measurements from these participants.
* Compare specific tissue sections from these participants with their excitation-emission matrices in order to identify the cell types contributing to the signal.

OUTLINE: Participants undergo placement of a fiber optic probe on one normal columnar cell site and one normal squamous cell site of the cervix during colposcopy*. The probe delivers laser light at a specific excitation wavelength and collects fluorescence from the entire emission wavelength range from the mucosa. Participants undergo biopsies of both sites.

NOTE: *The columnar epithelium will not be colposcopically visible in all patients, in which case 2 normal squamous sites will be measured

PROJECTED ACCRUAL: A total of 1,000 participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be individuals 18 years of age or older, who have voluntarily responded to advertisement in the form of posted flyers or word of mouth.
2. Subjects must sign an informed consent indicating awareness of the investigational nature of this study.

Exclusion Criteria:

1) Pregnant individuals will be ineligible for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1070 (Actual)
Dates: Start 1998-04; Primary Completion 2007-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Fluorescent Measurements of Cervix | Participation complete after readings of several 2.5 minutes fluorescent measurements and biopsies taken during colposcopy.
  Two fluorescent measurements of cervix, approximately 2.5 minutes each: 1)colposcopically normal columnar site, and 2) a colposcopically normal squamous site.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Rhodes, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org